CLINICAL TRIAL: NCT07073482
Title: Evaluating the Role of Stress Ball Use in Reducing Anxiety and Pain and Promoting Breastfeeding Following Elective Cesarean Section
Brief Title: Stress Ball Intervention for Anxiety, Pain, and Breastfeeding Following Elective Cesarean Section
Acronym: Anxiety
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Hatice Kusderci, MD, Samsun University
Other Study IDs: GOKAEK-2024/16/13
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Caesarean Section; Anxiety; Breast Milk
Keywords: caesarean section; breast milk; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group S: Stress ball group
  Interventions: Other: Using stress ball
- group C: control group

INTERVENTIONS:
Other: Using stress ball — The participant will be told that the stress balls will be used for 15 minutes during the surgery, and the researcher will inform the participant when the 15 minutes are up and the patient will be asked to release the balls.
  Groups: group S

SUMMARY:
Although pregnancy and birth are physiological processes, they create a significant burden and stress for the female body. The pregnancy period can cause permanent psychological changes as well as physiological ones. In the pre-operative period, patients experience anxiety for many reasons. In addition to general concerns such as health and surgery-related concerns, uncertainty about the end, moving away from home and loved ones, and interruption of daily tasks, there are also anesthesia-related concerns such as not being able to wake up after surgery, feeling pain after surgery, and waking up during surgery. These concerns become even more severe during pregnancy. One of the factors that increases anxiety and depression in the post-natal period is the type of birth. Anxiety and depression may develop due to complications that may occur after a cesarean section, the possibility of a delay in breastfeeding the baby, and pain. Early detection of anxiety and depression and taking precautions are important in order to increase the mother's quality of life and comfort after a cesarean section and to reduce anxiety and worry. In studies conducted to reduce anxiety and depression after cesarean section, there are studies showing that non-pharmacological evidence-based practices such as reiki, acupressure, hand and foot massage, yoga, reflexology, aromatherapy, skin contact and nursing care protocol are effective. Another effective method for reducing anxiety and pain is the stress ball. A stress ball is a soft toy that is usually no larger than 7 cm, is worn on the hand and manipulated with the fingers to relieve stress and muscle tension or to work the muscles. The stress ball, which is one of the distraction methods, is an effective method for providing cognitive focus. It has been observed that the stress ball method is used to reduce patients' anxiety and pain. There is no study in the literature examining the effect of stress ball use on intraoperative and postoperative pain and anxiety in patients undergoing cesarean section and its effects on breastfeeding. For these reasons, our study will contribute to the literature.

DETAILED DESCRIPTION:
After a caesarean section, which is an abdominal surgery, gastrointestinal movements may slow down, nausea, vomiting, cramps, and respiratory dysfunction may occur due to manipulations during the surgery and opioid use. This may cause increased anxiety in women. Factors that cause increased anxiety in women after a caesarean section include being exposed to a surgical operation, as well as prolonged transition to oral feeding, late mobilization, increased risk of infection, and delayed mother-baby interaction and milk secretion. Pain, fatigue, anxiety, and depression experienced after birth may cause mothers to be reluctant to breastfeed and decrease milk production. Early detection of anxiety and depression that may occur after a caesarean section and taking precautions for these situations contribute to improving the mother's quality of life, reducing anxiety and worry, and maintaining an effective and efficient mother-baby relationship. We planned this study to examine the effects of stress ball application during caesarean surgery on patients' anxiety, pain, and breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2 pregnant women

Exclusion Criteria:

* Those with known psychiatric or mental disorders, those using sedative medications, those under the age of 18 or over the age of 45, and those who do not want to be included in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women who underwent cesarean section
Study Population: Pregnant women who underwent cesarean section
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Anxiety Scale (VAS-A) | postoperative 48 hours
  It consists of a 10 cm long horizontal line. The left side contains the labels "No anxiety/worry" and the right side contains the labels "I am very anxious/worry". The VAS value is determined by measuring the distance between the top of the scale and the marked point. As the patient's anxiety level approaches 10, it shows that his anxiety increases.
State Trait Anxiety Inventory -STAI-II | postoperative 48 hours
  This scale consists of two parts: STAI-I and STAI-II. The scale consists of 20 items. Items 1-20 in the scale measure anxiety in four options. The statements in STAI-II are scored as; Almost never=1, Sometimes=2, Often=3, Almost always=4.
  The lowest score on the scale is 20, the highest score is 80. As the score increases, the anxiety level also increases.

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA AKDENİZ, asst prof, Principal Investigator — SAMSUN UNİVERSITY
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No